CLINICAL TRIAL: NCT03719963
Title: Preoperative Variables Affecting Outcome Of Cochlear Implant
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nashwa Ameer Mahmoud Mesaed, principle investigator, Assiut University
Other Study IDs: 17200178I
Record Dates: First submitted 2018-06-02; First posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Speech Cortex Disorder
MeSH Terms: interventions — Cochlear Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cochlear implant: Cochlear implantation is a powerful tool for helping children with severe to profound sensorineural hearing loss to gain the ability to hear, and to achieve age appropriate communication skills. Evaluating the development of auditory, speech, language skills and the personality of implanted child is useful for the parent, the teacher, the therapist, and the subsequent rehabilitation progress
  Interventions: Device: Cochlear implant

INTERVENTIONS:
Device: Cochlear implant — Cochlear implant for hearing process by surgical intervention

SUMMARY:
Cochlear implants (CIs) represent one of the most important achievements of modern medicine as, for the first time in history, an electronic device is able to restore a lost sense - hearing. As of December 2012, approximately 324,200 cochlear implants have been implanted worldwide. In the United States, roughly 58,000 devices have been implanted in adults and 38,000 in children .

The aim of this study is to assess the factors affecting the audiological, speech and language outcomes achieved by the recipients of multi-channel cochlear implants.

DETAILED DESCRIPTION:
Cochlear implants (CIs) represent one of the most important achievements of modern medicine as, for the first time in history, an electronic device is able to restore a lost sense - hearing. As of December 2012, approximately 324,200 cochlear implants have been implanted worldwide. In the United States, roughly 58,000 devices have been implanted in adults and 38,000 in children .

Cochlear implantation is a powerful tool for helping children with severe to profound sensorineural hearing loss to gain the ability to hear, and to achieve age appropriate communication skills. Evaluating the development of auditory, speech, language skills and the personality of implanted child is useful for the parent, the teacher, the therapist, and the subsequent rehabilitation progress .

However the final outcome in pediatric implantation is yet not entirely predictable as there are a large number of factors which alone or in combination will decide the outcome of cochlear implantation.

Categorizing these determinants increases the ability of clinicians to offer educated preoperative prognosis and might potentially allow for manipulation of variables in an attempt to achieve the best possible outcome .

Before implantation, a trial period with appropriate amplification combined with intensive auditory training should be attempted to ensure that maximal benefit is achieved.

Several factors have been reported to have an impact on the ability of prelingually deaf children to develop oral language skills after cochlear implantation. The most important and consistently reported variable that influences the ability to use auditory-only communication is the age at which the child is implanted .

Communication mode after implantation has also been frequently reported to be a factor that contributes to final speech and language outcome, with oral-only communication producing speech and language results superior to those observed in children who use a combination of sign and spoken language (total communication).

The wide range of speech perception abilities exhibited by cochlear implant recipients may depend in part upon differences in the central auditory processing abilities of implant users. One way to assess central auditory function in these individuals is to measure speech evoked cortical potentials. In particular, measuring cortical potentials that reflect auditory discrimination may provide insight into the central mechanisms underlying speech perception .

Moreover, if those cortical potentials can be recorded from cochlear implant users, comparing the potentials to the responses measured in normal listeners should indicate whether the brain's response to speech mediated by a cochlear implant is similar to the brain's response to speech processed by a normal cochlea. From a theoretical standpoint, the presence of cortical potentials in cochlear implant users may provide a unique window to viewing the central auditory system.

Aim of the study:

The aim of this study is to assess the factors affecting the audiological, speech and language outcomes achieved by the recipients of multichannel cochlear implants.

ELIGIBILITY:
Inclusion Criteria:

* a) Children with bilateral severe to profound sensorineural hearing loss. b) Age less than 6 years at time of implantation. c) Prelingual deafness

Exclusion Criteria:

* Incomplete follow up.
* post lingual children
* children with special needs such as mental retardation or autism

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Age less than 6years at time of implantation with history of cochlear implant
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
speech cortical evoked potential | 1 year
  Intelligent hearing system is the name of the instrument that will be used,speech stimulus that will used,cortical p1 and N1 waves that will be detected which is the outcome that we need to measure

CONTACTS AND LOCATIONS:
Overall Officials: Assiut university Faculty of medicine, University, Study Chair — www.emro.who.int/unified-medical -dictionary.html

IPD SHARING:
Plan to Share IPD: Yes
yes i agree to share the research plan
Supporting Information: SAP, CSR
Time Frame: 9-2018 for 6 months
Access Criteria: yes a agree to accrss

REFERENCES:
- [Result] Holt RF, Svirsky MA. An exploratory look at pediatric cochlear implantation: is earliest always best? Ear Hear. 2008 Aug;29(4):492-511. doi: 10.1097/AUD.0b013e31816c409f. PMID 18382374